CLINICAL TRIAL: NCT03626545
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study Evaluating the Efficacy and Safety of Canakinumab in Combination With Docetaxel Versus Placebo in Combination With Docetaxel in Adult Subjects With Non-small Cell Lung Cancer (NSCLC) Previously Treated With PD-(L)1 Inhibitors and Platinum-based Chemotherapy (CANOPY 2)
Brief Title: Phase III Study Evaluating Efficacy and Safety of Canakinumab in Combination With Docetaxel in Adult Subjects With Non-small Cell Lung Cancers as a Second or Third Line Therapy
Acronym: CANOPY-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was early terminated due to the lack of efficacy of study treatment observed in the analysis of the primary endpoint of the randomized part
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885V2301; 2018-002480-26 (EudraCT Number)
Record Dates: First submitted 2018-07-25; First posted 2018-08-13 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Non-Small-Cell Lung
Keywords: ACZ885; canakinumab; docetaxel; NSCLC; Non Small Cell Lung Cancer; Carcinoma; IL-1β; PD-(L)1; CANOPY; CANOPY-2; second or third line therapy; PD-(L)1 inhibitors; platinum-based chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Neoplasm Metastasis | interventions — canakinumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety run-in part: Canakinumab+docetaxel (Experimental): Participants were treated with full doses of docetaxel 75mg/m^2 intravenous and canakinumab 200 mg subcutaneous on Day 1 of each 21-Day cycle (dose level 1). Subjects were assessed for at least 2 complete cycles of treatment (21 days per cycle; a total of 42 days) for safety evaluation (DLT) to define RP3R. De-escalation to canakinumab 200 mg subcutaneous every 6 weeks + docetaxel 75 mg/m^2, every 3 weeks could also be considered.
  Interventions: Drug: Canakinumab; Drug: Docetaxel
- Randomized part: Canakinumab + docetaxel (Experimental): Participants were treated with canakinumab subcutaneous at RP3R and docetaxel at 75 mg/m^2 every 3 weeks
  Interventions: Drug: Canakinumab; Drug: Docetaxel
- Randomized part: Placebo + docetaxel (Placebo Comparator): Participants were treated with placebo subcutaneous at RP3R and docetaxel at 75 mg/m^2 every 3 weeks
  Interventions: Drug: Docetaxel; Other: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumab, 200 mg, subcutaneous. The initial dose regimen was once every 3 weeks (on Day 1 of each 21-day cycle)
  Other Names: ACZ885
  Arms: Randomized part: Canakinumab + docetaxel; Safety run-in part: Canakinumab+docetaxel
Drug: Docetaxel — Docetaxel 75mg/m^2, intravenous, administered on Day 1 of each 21-day cycle
Other: Placebo — Placebo, sub-cutaneous, admnistered at the RP3R defined in Part 1-safety run-in.
  Arms: Randomized part: Placebo + docetaxel

SUMMARY:
This study was designed to evaluate the role of canakinumab in combination with docetaxel in subjects with advanced non-small cell lung cancer (NSCLC) previously treated with PD-(L)1 inhibitors and platinum-based chemotherapy.

DETAILED DESCRIPTION:
This was a multicenter, Phase III study designed to evaluate the efficacy and safety of canakinumab in combination with docetaxel versus placebo in combination with docetaxel, as second- or third-line treatment. The study included adult subjects with advanced NSCLC whose disease had progressed after prior treatment with a PD-(L)1 inhibitor. Subjects had also been pre-treated with platinum-based chemotherapy, either given together with PD-(L)1 inhibitor or sequentially.

The study consisted of 2 parts:

* Part 1: Safety run-in. This part was conducted to confirm the Recommended Phase 3 Regimen (RP3R) of the canakinumab and docetaxel combination. Participants were treated for at least 2 complete cycles of treatment (21 days per cycle) for safety evaluation (DLT-Dose Limiting Toxicities) to define RP3R. Participants from the safety run-in part were treated until any discontinuation criteria were met. After treatment discontinuation, all participants were followed for safety evaluations during the safety follow up period (up to 130 days). Additionally, subjects who discontinued study treatment without prior documented disease progression continued efficacy assessments in the efficacy follow-up phase irrespective of the start of new antineoplastic therapy and until documented progressive disease as per protocol. After the RP3R was determined, enrollment in this part was closed and additional participants were enrolled in the randomized part (part 2) of the study. Ongoing patients from the safety run-in part continued their treatment at the assigned dose level according to the dose and schedule for the safety run-in part.
* Part 2: Randomized part. The randomized, double-blind, placebo-controlled part of the study opened after confirmation of the RP3R for the combination of canakinumab and docetaxel. Participants from the randomized part were treated until any discontinuation criteria were met as per protocol. After treatment discontinuation, all participants were followed for safety evaluations during the safety follow up period (up to 130 days). Additionally, subjects who discontinued study treatment without prior documented disease progression continued efficacy assessments in the efficacy follow-up phase irrespective of the start of new antineoplastic therapy and until documented progressive disease as per protocol.

Based on the lack of efficacy observed in the primary analysis, Novartis decided to halt canakinumab/placebo treatment. Subjects continued to receive docetaxel if they were deriving clinical benefit as per investigator assessment until discontinuation

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed advanced (stage IIIB) or metastatic NSCLC.
* Subject had received one prior platinum-based chemotherapy and one prior PD-(L)1 inhibitor therapy for locally advanced or metastatic disease.
* Subject with ECOG performance status (PS) of 0 or 1.
* Subject with at least 1 evaluable (measurable or non-measurable) lesion by RECIST 1.1 in solid tumors criteria.

Key Exclusion Criteria:

* Subject who previously received docetaxel, canakinumab (or another IL-1β inhibitor), or any systemic therapy for their locally advanced or metastatic NSCLC other than one platinum-based chemotherapy and one prior PD-(L)1 inhibitor.
* Subject with EGFRor ALK positive tumor.
* History of severe hypersensitivity reaction to monoclonal antibodies, taxanes or excipients of docetaxel or canakinumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- United States (6):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Saint Luke's Hospital/Marion Bloch Neuroscience Institute Dept of Regulatory, Kansas City, Missouri
  - Montefiore Medical Center Albert Einstein College of Med, The Bronx, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute Univ of Utah ., Salt Lake City, Utah
- Argentina (5):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, La Rioja
  - Novartis Investigative Site, Santiago del Estero
- Australia (2):
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Shepparton, Victoria
- Belgium (5):
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Roeselare
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Itajaí, Santa Catarina
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Santiago, Chile
- China (2):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Shanghai
- Czechia (2):
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Ostrava Vitkovice
- Denmark (2):
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense C
- France (5):
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Strasbourg
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Ulm
- Greece (2):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Törökbálint, Pest County, Hungary
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (3):
  - Novartis Investigative Site, Lucca, LU
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Aviano, PN
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (2):
  - Novartis Investigative Site, Pushkin Saint Petersburg
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Paz-Ares L, Goto Y, Wan-Teck Lim D, Halmos B, Chul Cho B, Cobo M, Luis Gonzalez Larriba J, Zhou C, Demedts I, Atmaca A, Baka S, Mookerjee B, Portella S, Zhu Z, Wu J, Demanse D, Dharan B, Reck M. Canakinumab in combination with docetaxel compared with docetaxel alone for the treatment of advanced non-small cell lung cancer following platinum-based doublet chemotherapy and immunotherapy (CANOPY-2): A multicenter, randomized, double-blind, phase 3 trial. Lung Cancer. 2024 Mar;189:107451. doi: 10.1016/j.lungcan.2023.107451. Epub 2024 Jan 16. PMID 38354535
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Safety run-in (Part 1) was conducted in 6 centers across 4 countries and the Randomized part (Part 2) was conducted in 85 centers across 26 countries.
Pre-assignment Details: In the randomized part, a total of 352 subjects were screened. 237 subjects completed the screening phase and were randomized in a 1:1 ratio to treatment with either canakinumab plus docetaxel or placebo plus docetaxel. Three randomized subjects in the placebo plus docetaxel group were not treated
Groups:
- Safety run-in Part: Canakinumab+Docetaxel: Participants were treated with full doses of docetaxel 75mg/m^2 intravenous and canakinumab 200 mg subcutaneous on Day 1 of each 21-Day cycle (dose level 1).
- Randomized Part: Canakinumab + Docetaxel: Participants were randomized to receive canakinumab subcutaneous at RP3R and docetaxel at 75 mg/m^2 on Day 1 of each 21-Day cycle
- Randomized Part: Placebo + Docetaxel: Participants were randomized to receive placebo subcutaneous at RP3R and docetaxel at 75 mg/m^2 on Day 1 of each 21-Day cycle
Period: Overall Study
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Started | 8 | 120 | 117
Treated | 8 | 120 | 114
Completed | 0 | 0 | 0
Not Completed | 8 | 120 | 117
Not completed — Progressive disease | 3 | 82 | 85
Not completed — Adverse Event | 3 | 13 | 10
Not completed — Physician Decision | 1 | 18 | 14
Not completed — Subject Decision | 0 | 5 | 5
Not completed — Death | 1 | 1 | 1
Not completed — Protocol Deviation | 0 | 1 | 1
Not completed — Guardian Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel | Total
Number analyzed (Participants) | 8 | 120 | 117 | 245
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (4.19) | 63.4 (9.13) | 62.2 (10.05) | 62.6 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 38 | 32 | 72
  Male | 6 | 82 | 85 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 91 | 83 | 182
  Asian | 0 | 22 | 27 | 49
  Unknown | 0 | 4 | 7 | 11
  Black or African American | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety run-in Part: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: Percentage of participants with DLTs. A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 42 days of docetaxel and canakinumab treatment.
Time Frame: During the first 42 days of dosing
Population: Participants in the safety run-in part to whom study treatment was assigned, who received at least one dose of any study treatment (including incomplete infusion) and met the minimum exposure criterion and have sufficient safety evaluations, or experienced a DLT during the first 42 days of dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 7
Participants | 1

2. Primary Outcome: Randomized Part: Overall Survival (OS)
Description: OS is defined as the time from randomization to date of death due to any cause. The OS distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated for each treatment group. If a subject was not known to have died, then OS was censored at the latest date the subject was known to be alive (on or before the cut-off date).
Time Frame: From randomization until death or final analysis data cutoff date (08-Jan-2021) whichever comes first (up to approximately (approx.) 18 months)
Population: Full Analysis Set (FAS) in randomized part: All participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Months | 10.55 [8.15 to 12.39] | 11.30 [8.54 to 13.80]
Statistical Analysis 1: Comparison: Randomized Part: Canakinumab + Docetaxel vs Randomized Part: Placebo + Docetaxel; Test type: Superiority; p = 0.633, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.76 to 1.48] — Hazard ratio was estimated using a Cox Proportional Hazards regression model stratified by line of therapy and histology

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR), as per investigator's assessment by RECIST 1.1. The 95% confidence intervals (CIs) were computed using Clopper and Pearson method.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Through final analysis data cutoff date of 08-Jan-2021 (assessed up to approx. 10 months for the safety run-in part and 18 months for the randomized part)
Population: FAS in Safety run-in part: all participants to whom study treatment was assigned and who received at least one dose of any study treatment (including incomplete infusion) FAS in Randomized part: all participants to whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 8 | 120 | 117
Percentage of participants | 0.0 [NA to NA] — NA: Not estimable because no participants had best overall response of CR or PR | 15.0 [9.1 to 22.7] | 13.7 [8.0 to 21.3]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first documented response of CR or PR to date of first documented progression or death, by investigator's assessment according to RECIST 1.1 criteria. The DOR distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated for each treatment group.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first documented response of CR or PR to date of first documented progression, death or final analysis data cutoff date (08-Jan-2021) whichever comes first (up to approx. 10 months for the safety run-in and 18 months for the randomized)
Population: FAS in Safety run-in part: all participants to whom study treatment was assigned and who received at least one dose of any study treatment (including incomplete infusion) for whom best overall response is CR or PR FAS in Randomized part: all participants to whom study treatment was assigned by randomization for whom best overall response is CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 0 | 18 | 16
Months |  | 4.14 [2.89 to 11.17] | 5.42 [4.17 to NA] — Not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with CR or PR or with stable disease (SD) as per investigator assessment according to RECIST 1.1 criteria. The 95% CIs were computed using Clopper and Pearson method.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 8 | 120 | 117
Percentage of participants | 62.5 [24.5 to 91.5] | 65.8 [56.6 to 74.2] | 61.5 [52.1 to 70.4]

6. Secondary Outcome: Randomized Part: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of the first documented radiological progression by investigator assessment according to RECIST 1.1 response criteria or death due to any cause.
  The PFS distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated for each treatment group. If a participant did not have disease progression or die at the analysis cut-off date, PFS was censored at the date of last adequate tumor assessment.
Time Frame: From randomization until disease progression, death or final analysis data cutoff date (08-Jan-2021) whichever comes first (assessed up to approx. 18 months)
Population: FAS in Randomized part: All participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Months | 4.17 [2.96 to 5.42] | 4.21 [3.06 to 5.13]

7. Secondary Outcome: Randomized Part: Time to Response (TTR)
Description: TTR is defined as the time from the date of randomization to the date of first documented response of either CR or PR, by investigator's assessment according to RECIST 1.1 criteria. The TTR distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated for each treatment group. Subjects without a confirmed CR or PR at the time of the analysis cut-off date were censored at the study-maximum follow-up time for subjects with a PFS event (i.e., disease progression or death due to any cause), or at the date of the last adequate tumor assessment for subjects without a PFS event.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From randomization until first documented response or final analysis data cutoff date (08-Jan-2021) whichever comes first (up to approx. 18 months)
Population: FAS in Randomized part: All participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Months | NA [NA to NA] — NA: Not evaluable due to the low number of participants with events | NA [NA to NA] — NA: Not evaluable due to the low number of participants with events

8. Secondary Outcome: Randomized Part: Time to Definitive 10-point Deterioration (TTD) Symptom Scores of Chest Pain, Cough and Dyspnea Per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) Lung Cancer (LC13) Questionnaire
Description: The EORTC QLQ-LC13 comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, dyspnea, and chest pain) and treatment-related symptoms from conventional chemotherapy and radiotherapy (ie. hair loss, neuropathy, sore mouth, and dysphagia). Scores for each scale and single-item range from 0 to 100, with higher scores indicating higher level of symptoms. TTD for chest pain, cough and dyspnea is defined as the time from randomization to the date of event, which is defined as at least 10 points absolute worsening from baseline of the corresponding scale score, with no later change below this threshold ie.<10 points was observed or if this worsening was observed at the last assessment for the subject, or death due to any cause (whichever occurs earlier). If a subject did not have an event, TTD was censored at the last adequate assessment.
Time Frame: From baseline through final analysis data cutoff date of 08-Jan-2021 (assessed up to approx. 18 months)
Population: FAS in Randomized part: All participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Months
  Chest Pain | 7.23 [4.96 to NA] — NA: Upper limit was not reached due to the insufficient number of participants with events | 13.14 [7.06 to NA] — NA: Upper limit was not reached due to the insufficient number of participants with events
  Cough | 7.23 [5.09 to NA] — NA: Upper limit was not reached due to the insufficient number of participants with events | 13.14 [7.85 to NA] — NA: Upper limit was not reached due to the insufficient number of participants with events
  Dyspnea | 3.45 [2.14 to 4.83] | 4.27 [2.63 to 5.65]

9. Secondary Outcome: Randomized Part: Time to Definitive 10-point Deterioration in Global Health Status (GHS)/Quality of Life (QoL), Shortness of Breath and Pain Per EORTC QLQ-C30 Questionnaire
Description: The EORTC QLQ-C30 includes 5 functional scales (physical,role,cognitive,emotional and social), 3 symptom scales (fatigue,pain and nausea/vomiting), a GHS/QoL scale, and 6 single items (constipation,diarrhea,insomnia,shortness of breath,appetite loss and financial difficulties). For each scale and single-item, scores range between 0 and 100. A high score for functional scales/ GHS/QoL represents better functioning or QoL, a high score for symptom scales/single items represents significant symptomatology. TTD in GHS/QoL, shortness of breath and pain is defined as the time from randomization to the date of event, defined as at least 10 points absolute worsening from baseline of the corresponding scale score, with no later change below this threshold i.e.<10 points was observed or if this worsening was observed at the last assessment for the subject, or death due to any cause (whichever occurs earlier). If a subject did not have an event, TTD was censored at the last adequate assessment.
Time Frame: From baseline through final analysis data cutoff date of 08-Jan-2021 (assessed up to approx. 18 months)
Population: FAS in Randomized part: All participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Months
  GHS/QOL | 4.83 [3.48 to 6.97] | 7.16 [4.80 to 13.14]
  Shortness of breath | 6.57 [4.60 to 7.89] | 5.78 [4.27 to NA] — NA: Upper limit was not reached due to the insufficient number of participants with events
  Pain | 6.05 [4.47 to 7.72] | 8.54 [4.27 to 10.38]

10. Secondary Outcome: Randomized Part: Change From Baseline in GHS/QoL, Shortness of Breath and Pain Scores as Per the EORTC QLQ C30 Questionnaire
Description: The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and 6 single items (constipation, diarrhea, insomnia, dyspnoea, appetite loss and financial difficulties). For each scale and item, scores range 0-100. A high score for functional scales/QoL represents better functioning/QoL; a high score for symptom scales and items represents significant symptomatology. Changes from baseline in QoL, shortness of breath and pain scores are presented. For QoL, a negative change from baseline indicates improvement; for shortness of breath and pain a positive change from baseline indicates improvement. For subjects who discontinued treatment without disease progression, post-treatment efficacy visits 1, 2, 3 and 5 were conducted every 6 weeks (for the first 12 months since start of treatment) and every 12 weeks (after 12 months since start of treatment) until disease progression
Time Frame: Baseline, every 3 weeks from Week 3 until end of treatment, every 6 or 12 weeks post-treatment until progression (post-treatment efficacy visits), 7 and 28 days post progression through final analysis cutoff date of 08Jan2021 (up to approx. 18 months)
Population: FAS in Randomized part: All participants to whom study treatment was assigned by randomization. Number analyzed represents participants with data available at the specified data points
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Score on a scale
  GHS/QoL: Week 3: number analyzed (Participants) | 92 | 103
  GHS/QoL: Week 3 | -0.5 (18.34) | 1.8 (21.51)
  GHS/QoL: Week 6: number analyzed (Participants) | 78 | 85
  GHS/QoL: Week 6 | -3.3 (17.48) | 1.4 (22.19)
  GHS/QoL: Week 9: number analyzed (Participants) | 65 | 70
  GHS/QoL: Week 9 | -2.7 (20.04) | -0.4 (23.50)
  GHS/QoL: Week 12: number analyzed (Participants) | 63 | 60
  GHS/QoL: Week 12 | -7.4 (19.75) | 2.5 (22.14)
  GHS/QoL: Week 15: number analyzed (Participants) | 51 | 50
  GHS/QoL: Week 15 | -2.9 (19.85) | -4.2 (22.60)
  GHS/QoL: Week 18: number analyzed (Participants) | 51 | 48
  GHS/QoL: Week 18 | -3.9 (22.75) | 2.8 (24.69)
  GHS/QoL: Week 21: number analyzed (Participants) | 40 | 38
  GHS/QoL: Week 21 | -3.5 (25.31) | -4.2 (27.25)
  GHS/QoL: Week 24: number analyzed (Participants) | 35 | 34
  GHS/QoL: Week 24 | -3.6 (16.08) | -0.7 (24.90)
  GHS/QoL: Week 27: number analyzed (Participants) | 23 | 27
  GHS/QoL: Week 27 | -4.7 (16.25) | -2.2 (26.51)
  GHS/QoL: Week 30: number analyzed (Participants) | 18 | 25
  GHS/QoL: Week 30 | -3.7 (19.43) | -5.7 (30.31)
  GHS/QoL: Week 33: number analyzed (Participants) | 13 | 20
  GHS/QoL: Week 33 | -3.2 (15.79) | 0.4 (31.82)
  GHS/QoL: Week 36: number analyzed (Participants) | 11 | 15
  GHS/QoL: Week 36 | -4.5 (15.97) | 3.3 (27.06)
  GHS/QoL: Week 39: number analyzed (Participants) | 10 | 14
  GHS/QoL: Week 39 | -5.8 (18.02) | 1.2 (28.28)
  GHS/QoL: Week 42: number analyzed (Participants) | 10 | 15
  GHS/QoL: Week 42 | -9.2 (16.41) | 2.8 (29.15)
  GHS/QoL: Week 45: number analyzed (Participants) | 7 | 12
  GHS/QoL: Week 45 | -3.6 (16.57) | -3.5 (22.32)
  GHS/QoL: Week 48: number analyzed (Participants) | 6 | 9
  GHS/QoL: Week 48 | -8.3 (19.72) | -13.9 (13.82)
  GHS/QoL: Week 51: number analyzed (Participants) | 6 | 10
  GHS/QoL: Week 51 | -8.3 (16.67) | -6.7 (21.80)
  GHS/QoL: Week 54: number analyzed (Participants) | 6 | 7
  GHS/QoL: Week 54 | -6.9 (17.01) | -4.8 (31.86)
  GHS/QoL: Week 57: number analyzed (Participants) | 4 | 5
  GHS/QoL: Week 57 | -12.5 (14.43) | -8.3 (36.32)
  GHS/QoL: Week 60: number analyzed (Participants) | 3 | 4
  GHS/QoL: Week 60 | -8.3 (22.05) | 2.1 (38.71)
  GHS/QoL: Week 63: number analyzed (Participants) | 3 | 3
  GHS/QoL: Week 63 | -5.6 (17.35) | 2.8 (4.81)
  GHS/QoL: Week 66: number analyzed (Participants) | 2 | 2
  GHS/QoL: Week 66 | 8.3 (11.79) | -8.3 (11.79)
  GHS/QoL: Week 69: number analyzed (Participants) | 1 | 2
  GHS/QoL: Week 69 | 16.7 (NA) — NA: The standard deviation was not estimable as there was only one participant. | 0.0 (23.57)
  GHS/QoL: Week 72: number analyzed (Participants) | 0 | 2
  GHS/QoL: Week 72 |  | -8.3 (11.79)
  GHS/QoL: Week 75: number analyzed (Participants) | 0 | 1
  GHS/QoL: Week 75 |  | -16.7 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  GHS/QoL: Week 78: number analyzed (Participants) | 0 | 1
  GHS/QoL: Week 78 |  | -16.7 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  GHS/QoL: post treatment efficacy visit 1: number analyzed (Participants) | 2 | 3
  GHS/QoL: post treatment efficacy visit 1 | -16.7 (11.79) | 5.6 (9.62)
  GHS/QoL: post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  GHS/QoL: post treatment efficacy visit 2 | -16.7 (16.67) | 16.7 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  GHS/QoL: post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  GHS/QoL: post treatment efficacy visit 3 |  | -8.3 (23.57)
  GHS/QoL: post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  GHS/QoL: post treatment efficacy visit 5 |  | 25.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  GHS/QoL: 7 days post disease progression: number analyzed (Participants) | 31 | 29
  GHS/QoL: 7 days post disease progression | -7.5 (26.65) | -4.6 (22.11)
  GHS/QoL: 28 days post disease progression: number analyzed (Participants) | 18 | 17
  GHS/QoL: 28 days post disease progression | -3.7 (29.60) | -7.8 (20.08)
  Shortness of breath: Week 3: number analyzed (Participants) | 92 | 103
  Shortness of breath: Week 3 | 31.2 (28.30) | 31.7 (30.02)
  Shortness of breath: Week 6: number analyzed (Participants) | 78 | 84
  Shortness of breath: Week 6 | 7.3 (24.99) | 4.0 (28.06)
  Shortness of breath: Week 9: number analyzed (Participants) | 65 | 70
  Shortness of breath: Week 9 | 6.7 (27.13) | 5.7 (28.36)
  Shortness of breath: Week 12: number analyzed (Participants) | 63 | 60
  Shortness of breath: Week 12 | 12.2 (25.61) | 4.4 (29.73)
  Shortness of breath: Week 15: number analyzed (Participants) | 51 | 50
  Shortness of breath: Week 15 | 7.8 (21.69) | 7.3 (29.58)
  Shortness of breath: Week 18: number analyzed (Participants) | 51 | 48
  Shortness of breath: Week 18 | 8.5 (26.54) | 3.5 (30.93)
  Shortness of breath: Week 21: number analyzed (Participants) | 40 | 38
  Shortness of breath: Week 21 | 34.2 (29.71) | 29.8 (27.72)
  Shortness of breath: Week 24: number analyzed (Participants) | 35 | 34
  Shortness of breath: Week 24 | 4.8 (21.61) | 6.9 (32.60)
  Shortness of breath: Week 27: number analyzed (Participants) | 23 | 27
  Shortness of breath: Week 27 | 13.0 (24.08) | -1.2 (36.38)
  Shortness of breath: Week 30: number analyzed (Participants) | 18 | 25
  Shortness of breath: Week 30 | 16.7 (20.61) | 5.3 (38.10)
  Shortness of breath: Week 33: number analyzed (Participants) | 13 | 20
  Shortness of breath: Week 33 | 17.9 (22.01) | -1.7 (39.70)
  Shortness of breath: Week 36: number analyzed (Participants) | 11 | 15
  Shortness of breath: Week 36 | 9.1 (21.56) | -2.2 (32.04)
  Shortness of breath: Week 39: number analyzed (Participants) | 10 | 14
  Shortness of breath: Week 39 | 33.3 (27.22) | 40.5 (26.73)
  Shortness of breath: Week 42: number analyzed (Participants) | 10 | 15
  Shortness of breath: Week 42 | 23.3 (27.44) | -6.7 (31.37)
  Shortness of breath: Week 45: number analyzed (Participants) | 7 | 12
  Shortness of breath: Week 45 | 9.5 (31.71) | 8.3 (40.51)
  Shortness of breath: Week 48: number analyzed (Participants) | 6 | 9
  Shortness of breath: Week 48 | 22.2 (34.43) | 3.7 (26.06)
  Shortness of breath: Week 51: number analyzed (Participants) | 6 | 10
  Shortness of breath: Week 51 | 16.7 (18.26) | 0.0 (22.22)
  Shortness of breath: Week 54: number analyzed (Participants) | 6 | 7
  Shortness of breath: Week 54 | 11.1 (17.21) | 9.5 (37.09)
  Shortness of breath: Week 57: number analyzed (Participants) | 4 | 5
  Shortness of breath: Week 57 | 8.3 (31.91) | 20.0 (38.01)
  Shortness of breath: Week 60: number analyzed (Participants) | 3 | 4
  Shortness of breath: Week 60 | 0.0 (33.33) | 16.7 (43.03)
  Shortness of breath: Week 63: number analyzed (Participants) | 3 | 3
  Shortness of breath: Week 63 | 0.0 (33.33) | 0.0 (33.33)
  Shortness of breath: Week 66: number analyzed (Participants) | 2 | 2
  Shortness of breath: Week 66 | -16.7 (23.57) | 0.0 (47.14)
  Shortness of breath: Week 69: number analyzed (Participants) | 1 | 2
  Shortness of breath: Week 69 | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. | -16.7 (70.71)
  Shortness of breath: Week 72: number analyzed (Participants) | 0 | 2
  Shortness of breath: Week 72 |  | -16.7 (70.71)
  Shortness of breath: Week 75: number analyzed (Participants) | 0 | 1
  Shortness of breath: Week 75 |  | 33.3 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Shortness of breath: Week 78: number analyzed (Participants) | 0 | 1
  Shortness of breath: Week 78 |  | 33.3 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Shortness of breath: post treatment efficacy visit 1: number analyzed (Participants) | 2 | 3
  Shortness of breath: post treatment efficacy visit 1 | 33.3 (47.14) | 33.3 (33.33)
  Shortness of breath: post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  Shortness of breath: post treatment efficacy visit 2 | 0.0 (33.33) | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Shortness of breath: post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  Shortness of breath: post treatment efficacy visit 3 |  | 16.7 (23.57)
  Shortness of breath: post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  Shortness of breath: post treatment efficacy visit 5 |  | 0.00 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Shortness of breath: 7 days post disease progression: number analyzed (Participants) | 31 | 29
  Shortness of breath: 7 days post disease progression | 8.6 (21.03) | 8.0 (29.08)
  Shortness of breath: 28 days post disease progression: number analyzed (Participants) | 18 | 17
  Shortness of breath: 28 days post disease progression | 3.7 (27.75) | 15.7 (29.15)
  Pain: Week 3: number analyzed (Participants) | 92 | 102
  Pain: Week 3 | -5.1 (21.07) | -2.0 (22.53)
  Pain: Week 6: number analyzed (Participants) | 78 | 85
  Pain: Week 6 | -5.1 (20.33) | -1.6 (24.07)
  Pain: Week 9: number analyzed (Participants) | 65 | 70
  Pain: Week 9 | -4.1 (19.33) | -3.1 (21.85)
  Pain: Week 12: number analyzed (Participants) | 62 | 60
  Pain: Week 12 | 2.2 (24.61) | -1.4 (27.32)
  Pain: Week 15: number analyzed (Participants) | 51 | 50
  Pain: Week 15 | -0.7 (20.81) | 0.7 (22.07)
  Pain: Week 18: number analyzed (Participants) | 51 | 48
  Pain: Week 18 | 2.3 (23.34) | 0.7 (25.25)
  Pain: Week 21: number analyzed (Participants) | 40 | 38
  Pain: Week 21 | 3.3 (24.52) | 0.0 (25.70)
  Pain: Week 24: number analyzed (Participants) | 35 | 34
  Pain: Week 24 | 25.2 (25.36) | 19.1 (21.76)
  Pain: Week 27: number analyzed (Participants) | 23 | 27
  Pain: Week 27 | 1.4 (22.42) | 1.2 (19.57)
  Pain: Week 30: number analyzed (Participants) | 18 | 25
  Pain: Week 30 | 2.8 (19.17) | 4.0 (26.03)
  Pain: Week 33: number analyzed (Participants) | 12 | 20
  Pain: Week 33 | -8.3 (19.46) | 6.7 (21.22)
  Pain: Week 36: number analyzed (Participants) | 11 | 15
  Pain: Week 36 | 22.7 (17.12) | 26.7 (23.40)
  Pain: Week 39: number analyzed (Participants) | 10 | 14
  Pain: Week 39 | -10.0 (21.08) | 10.7 (31.08)
  Pain: Week 42: number analyzed (Participants) | 10 | 15
  Pain: Week 42 | -3.3 (10.54) | 11.1 (30.65)
  Pain: Week 45: number analyzed (Participants) | 7 | 12
  Pain: Week 45 | -11.9 (23.00) | 15.3 (30.53)
  Pain: Week 48: number analyzed (Participants) | 6 | 9
  Pain: Week 48 | -5.6 (22.77) | 5.6 (20.41)
  Pain: Week 51: number analyzed (Participants) | 6 | 10
  Pain: Week 51 | 2.8 (24.53) | 8.3 (18.00)
  Pain: Week 54: number analyzed (Participants) | 6 | 7
  Pain: Week 54 | 8.3 (20.41) | -2.4 (32.53)
  Pain: Week 57: number analyzed (Participants) | 4 | 5
  Pain: Week 57 | 0.0 (13.61) | 6.7 (19.00)
  Pain: Week 60: number analyzed (Participants) | 3 | 4
  Pain: Week 60 | 16.7 (16.67) | 0.0 (36.00)
  Pain: Week 63: number analyzed (Participants) | 3 | 3
  Pain: Week 63 | 5.6 (25.46) | -16.7 (16.7)
  Pain: Week 66: number analyzed (Participants) | 2 | 2
  Pain: Week 66 | 0.0 (0.00) | 0.0 (0.00)
  Pain: Week 69: number analyzed (Participants) | 1 | 2
  Pain: Week 69 | 33.3 (NA) — NA: The standard deviation was not estimable as there was only one participant. | 8.3 (11.79)
  Pain: Week 72: number analyzed (Participants) | 0 | 2
  Pain: Week 72 |  | 0.0 (0.00)
  Pain: Week 75: number analyzed (Participants) | 0 | 1
  Pain: Week 75 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Pain: Week 78: number analyzed (Participants) | 0 | 1
  Pain: Week 78 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Pain: post treatment efficacy visit 1: number analyzed (Participants) | 2 | 3
  Pain: post treatment efficacy visit 1 | -33.3 (23.57) | -11.1 (19.25)
  Pain: post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  Pain: post treatment efficacy visit 2 | 0.0 (16.67) | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Pain: post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  Pain: post treatment efficacy visit 3 |  | 33.3 (0.00)
  Pain: post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  Pain: post treatment efficacy visit 5 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Pain: 7 days post disease progression: number analyzed (Participants) | 31 | 29
  Pain: 7 days post disease progression | 1.6 (18.44) | 2.3 (31.41)
  Pain: 28 days post disease progression: number analyzed (Participants) | 18 | 17
  Pain: 28 days post disease progression | 9.3 (23.02) | 13.7 (20.61)

11. Secondary Outcome: Randomized Part: Change From Baseline in Chest Pain, Cough and Dyspnea Scores as Per the EORTC-QLQ LC13 Questionnaire
Description: The EORTC QLQ-LC13 is a 13-item questionnaire. It comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, dyspnea, and chest pain) and treatment-related symptoms from conventional chemotherapy and radiotherapy (ie, hair loss, neuropathy, sore mouth, and dysphagia). Scores for each scale and single-item range from 0 to 100, with higher scores indicating higher ("worse") level of symptoms. Changes from baseline in chest pain, cough and dyspnea scores are presented. A positive change from baseline indicates improvement. For subjects who discontinued treatment without disease progression, post-treatment efficacy visits 1, 2, 3 and 5 were conducted every 6 weeks (for the first 12 months since start of treatment) and every 12 weeks (after 12 months since start of treatment) until disease progression
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Score on a scale
  Chest pain: Week 3: number analyzed (Participants) | 92 | 102
  Chest pain: Week 3 | -2.2 (16.24) | -3.2 (24.48)
  Chest pain: Week 6: number analyzed (Participants) | 78 | 85
  Chest pain: Week 6 | 0.4 (19.73) | -3.9 (24.89)
  Chest pain: Week 9: number analyzed (Participants) | 65 | 70
  Chest pain: Week 9 | 0.5 (19.09) | -3.8 (22.37)
  Chest pain: Week 12: number analyzed (Participants) | 63 | 60
  Chest pain: Week 12 | 1.1 (23.16) | -3.3 (24.32)
  Chest pain: Week 15: number analyzed (Participants) | 51 | 49
  Chest pain: Week 15 | 0.7 (25.38) | -0.7 (24.05)
  Chest pain: Week 18: number analyzed (Participants) | 51 | 49
  Chest pain: Week 18 | 0.7 (21.59) | -4.1 (26.90)
  Chest pain: Week 21: number analyzed (Participants) | 40 | 38
  Chest pain: Week 21 | 2.5 (26.57) | 0.9 (18.15)
  Chest pain: Week 24: number analyzed (Participants) | 35 | 34
  Chest pain: Week 24 | 1.9 (21.30) | -1.0 (17.38)
  Chest pain: Week 27: number analyzed (Participants) | 23 | 27
  Chest pain: Week 27 | 2.9 (19.88) | 6.2 (27.79)
  Chest pain: Week 30: number analyzed (Participants) | 18 | 25
  Chest pain: Week 30 | 3.7 (19.43) | 6.7 (23.57)
  Chest pain: Week 33: number analyzed (Participants) | 13 | 19
  Chest pain: Week 33 | -5.1 (18.49) | 0.0 (15.71)
  Chest pain: Week 36: number analyzed (Participants) | 11 | 15
  Chest pain: Week 36 | -9.1 (15.57) | 0.0 (21.82)
  Chest pain: Week 39: number analyzed (Participants) | 10 | 14
  Chest pain: Week 39 | 0.0 (22.22) | 9.5 (30.46)
  Chest pain: Week 42: number analyzed (Participants) | 10 | 15
  Chest pain: Week 42 | 0.0 (15.71) | 0.0 (17.82)
  Chest pain: Week 45: number analyzed (Participants) | 7 | 12
  Chest pain: Week 45 | 0.0 (19.25) | 8.3 (15.08)
  Chest pain: Week 48: number analyzed (Participants) | 6 | 9
  Chest pain: Week 48 | 0.0 (21.08) | 11.1 (16.67)
  Chest pain: Week 51: number analyzed (Participants) | 6 | 10
  Chest pain: Week 51 | 0.0 (21.08) | 10.0 (22.50)
  Chest pain: Week 54: number analyzed (Participants) | 6 | 7
  Chest pain: Week 54 | 0.0 (21.08) | 9.5 (31.71)
  Chest pain: Week 57: number analyzed (Participants) | 4 | 5
  Chest pain: Week 57 | 0.0 (0.00) | 20.0 (18.26)
  Chest pain: Week 60: number analyzed (Participants) | 3 | 4
  Chest pain: Week 60 | -11.1 (19.25) | 25.0 (16.67)
  Chest pain: Week 63: number analyzed (Participants) | 3 | 3
  Chest pain: Week 63 | 0.0 (33.33) | 0.0 (0.00)
  Chest pain: Week 66: number analyzed (Participants) | 2 | 2
  Chest pain: Week 66 | 0.0 (47.14) | 0.0 (0.00)
  Chest pain: Week 69: number analyzed (Participants) | 1 | 2
  Chest pain: Week 69 | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. | 0.0 (0.00)
  Chest pain: Week 72: number analyzed (Participants) | 0 | 2
  Chest pain: Week 72 |  | 0.0 (0.00)
  Chest pain: Week 75: number analyzed (Participants) | 0 | 1
  Chest pain: Week 75 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Chest pain: Week 78: number analyzed (Participants) | 0 | 1
  Chest pain: Week 78 |  | 33.3 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Chest pain:Post treatment efficacy visit 1: number analyzed (Participants) | 2 | 3
  Chest pain:Post treatment efficacy visit 1 | 0.0 (0.00) | -22.2 (19.25)
  Chest pain: Post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  Chest pain: Post treatment efficacy visit 2 | 11.1 (19.25) | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Chest pain: Post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  Chest pain: Post treatment efficacy visit 3 |  | 16.7 (23.57)
  Chest pain: Post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  Chest pain: Post treatment efficacy visit 5 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Chest pain: 7 days post disease progression: number analyzed (Participants) | 31 | 29
  Chest pain: 7 days post disease progression | 5.4 (17.42) | -5.7 (21.95)
  Chest pain: 28 days post disease progression: number analyzed (Participants) | 18 | 16
  Chest pain: 28 days post disease progression | 14.8 (26.13) | -2.1 (25.73)
  Coughing: Week 3: number analyzed (Participants) | 92 | 103
  Coughing: Week 3 | 0.0 (21.54) | -3.2 (24.03)
  Coughing: Week 6: number analyzed (Participants) | 78 | 85
  Coughing: Week 6 | 3.0 (26.42) | -4.7 (27.77)
  Coughing: Week 9: number analyzed (Participants) | 65 | 70
  Coughing: Week 9 | 2.6 (32.44) | 0.5 (25.69)
  Coughing: Week 12: number analyzed (Participants) | 63 | 60
  Coughing: Week 12 | 4.8 (33.79) | 0.0 (26.75)
  Coughing: Week 15: number analyzed (Participants) | 51 | 49
  Coughing: Week 15 | 2.0 (27.82) | -0.7 (24.05)
  Coughing: Week 18: number analyzed (Participants) | 51 | 49
  Coughing: Week 18 | -1.3 (26.63) | 0.0 (31.18)
  Coughing: Week 21: number analyzed (Participants) | 40 | 38
  Coughing: Week 21 | -4.2 (30.37) | -4.4 (28.13)
  Coughing: Week 24: number analyzed (Participants) | 35 | 34
  Coughing: Week 24 | -1.0 (31.81) | -3.9 (24.29)
  Coughing: Week 27: number analyzed (Participants) | 23 | 27
  Coughing: Week 27 | -4.3 (25.23) | -1.2 (28.47)
  Coughing: Week 30: number analyzed (Participants) | 18 | 25
  Coughing: Week 30 | -5.6 (36.60) | -4.0 (26.03)
  Coughing: Week 33: number analyzed (Participants) | 13 | 19
  Coughing: Week 33 | 2.6 (16.45) | -3.5 (26.98)
  Coughing: Week 36: number analyzed (Participants) | 11 | 15
  Coughing: Week 36 | 12.1 (16.82) | -6.7 (28.73)
  Coughing: Week 39: number analyzed (Participants) | 10 | 14
  Coughing: Week 39 | 3.3 (18.92) | -4.8 (25.68)
  Coughing: Week 42: number analyzed (Participants) | 10 | 15
  Coughing: Week 42 | 6.7 (26.29) | -8.9 (29.46)
  Coughing: Week 45: number analyzed (Participants) | 7 | 12
  Coughing: Week 45 | 0.0 (19.25) | 2.8 (17.16)
  Coughing: Week 48: number analyzed (Participants) | 6 | 9
  Coughing: Week 48 | 11.1 (17.21) | 3.7 (20.03)
  Coughing: Week 51: number analyzed (Participants) | 6 | 10
  Coughing: Week 51 | 16.7 (18.26) | -3.3 (18.92)
  Coughing: Week 54: number analyzed (Participants) | 6 | 7
  Coughing: Week 54 | 16.7 (18.26) | -4.8 (23.00)
  Coughing: Week 57: number analyzed (Participants) | 4 | 5
  Coughing: Week 57 | -8.3 (16.67) | 6.7 (27.89)
  Coughing: Week 60: number analyzed (Participants) | 3 | 4
  Coughing: Week 60 | 0.0 (0.00) | -8.3 (31.91)
  Coughing: Week 63: number analyzed (Participants) | 3 | 3
  Coughing: Week 63 | 0.0 (0.00) | -11.1 (19.25)
  Coughing: Week 66: number analyzed (Participants) | 2 | 2
  Coughing: Week 66 | -16.7 (23.57) | -16.7 (23.57)
  Coughing: Week 69: number analyzed (Participants) | 1 | 2
  Coughing: Week 69 | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. | -33.3 (47.14)
  Coughing: Week 72: number analyzed (Participants) | 0 | 2
  Coughing: Week 72 |  | -33.3 (47.14)
  Coughing: Week 75: number analyzed (Participants) | 0 | 1
  Coughing: Week 75 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Coughing: Week 78: number analyzed (Participants) | 0 | 1
  Coughing: Week 78 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Coughing: Post treatment efficacy visit 1: number analyzed (Participants) | 2 | 3
  Coughing: Post treatment efficacy visit 1 | 0.0 (0.00) | 0.0 (0.00)
  Coughing: Post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  Coughing: Post treatment efficacy visit 2 | -22.2 (19.25) | 33.3 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Coughing: Post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  Coughing: Post treatment efficacy visit 3 |  | -16.7 (23.57)
  Coughing: Post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  Coughing: Post treatment efficacy visit 5 |  | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Coughing: 7 days post disease progression: number analyzed (Participants) | 31 | 29
  Coughing: 7 days post disease progression | -1.1 (25.07) | 3.4 (31.30)
  Coughing: 28 days post disease progression: number analyzed (Participants) | 18 | 16
  Coughing: 28 days post disease progression | -3.7 (27.75) | -4.2 (31.91)
  Dyspnea: Week 3: number analyzed (Participants) | 92 | 103
  Dyspnea: Week 3 | 4.8 (17.84) | 2.9 (18.47)
  Dyspnea: Week 6: number analyzed (Participants) | 78 | 85
  Dyspnea: Week 6 | 4.4 (16.83) | 5.0 (19.59)
  Dyspnea: Week 9: number analyzed (Participants) | 65 | 70
  Dyspnea: Week 9 | 4.8 (19.44) | 5.2 (20.17)
  Dyspnea: Week 12: number analyzed (Participants) | 63 | 60
  Dyspnea: Week 12 | 7.4 (19.25) | 6.9 (20.57)
  Dyspnea: Week 15: number analyzed (Participants) | 51 | 49
  Dyspnea: Week 15 | 6.5 (16.66) | 10.9 (21.69)
  Dyspnea: Week 18: number analyzed (Participants) | 51 | 49
  Dyspnea: Week 18 | 10.2 (19.98) | 4.3 (22.43)
  Dyspnea: Week 21: number analyzed (Participants) | 40 | 38
  Dyspnea: Week 21 | 8.9 (19.36) | 6.7 (21.07)
  Dyspnea: Week 24: number analyzed (Participants) | 35 | 34
  Dyspnea: Week 24 | 7.9 (23.89) | 9.2 (20.19)
  Dyspnea: Week 27: number analyzed (Participants) | 23 | 27
  Dyspnea: Week 27 | 10.1 (21.43) | 8.6 (20.52)
  Dyspnea: Week 30: number analyzed (Participants) | 18 | 25
  Dyspnea: Week 30 | 8.0 (14.66) | 8.0 (21.40)
  Dyspnea: Week 33: number analyzed (Participants) | 13 | 19
  Dyspnea: Week 33 | 13.7 (17.66) | 7.0 (22.89)
  Dyspnea: Week 36: number analyzed (Participants) | 11 | 15
  Dyspnea: Week 36 | 12.1 (22.47) | 7.4 (21.28)
  Dyspnea: Week 39: number analyzed (Participants) | 10 | 14
  Dyspnea: Week 39 | 14.4 (16.60) | 10.3 (25.21)
  Dyspnea: Week 42: number analyzed (Participants) | 10 | 15
  Dyspnea: Week 42 | 20.0 (27.62) | 3.0 (23.18)
  Dyspnea: Week 45: number analyzed (Participants) | 7 | 12
  Dyspnea: Week 45 | 20.6 (26.00) | 13.0 (20.56)
  Dyspnea: Week 48: number analyzed (Participants) | 6 | 9
  Dyspnea: Week 48 | 20.4 (30.97) | 14.8 (13.61)
  Dyspnea: Week 51: number analyzed (Participants) | 6 | 10
  Dyspnea: Week 51 | 22.2 (29.81) | 7.8 (15.76)
  Dyspnea: Week 54: number analyzed (Participants) | 6 | 7
  Dyspnea: Week 54 | 22.2 (26.29) | 12.7 (13.50)
  Dyspnea: Week 57: number analyzed (Participants) | 4 | 5
  Dyspnea: Week 57 | 19.4 (31.91) | 11.1 (11.11)
  Dyspnea: Week 60: number analyzed (Participants) | 3 | 4
  Dyspnea: Week 60 | 25.9 (44.91) | -2.8 (24.64)
  Dyspnea: Week 63: number analyzed (Participants) | 3 | 3
  Dyspnea: Week 63 | 18.5 (44.91) | -3.7 (12.83)
  Dyspnea: Week 66: number analyzed (Participants) | 2 | 2
  Dyspnea: Week 66 | -11.1 (15.71) | 0.0 (15.71)
  Dyspnea: Week 69: number analyzed (Participants) | 1 | 2
  Dyspnea: Week 69 | -22.2 (NA) — NA: The standard deviation was not estimable as there was only one participant. | -11.1 (47.14)
  Dyspnea: Week 72: number analyzed (Participants) | 0 | 2
  Dyspnea: Week 72 |  | -11.1 (47.14)
  Dyspnea: Week 75: number analyzed (Participants) | 0 | 1
  Dyspnea: Week 75 |  | 22.2 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Dyspnea: Week 78: number analyzed (Participants) | 0 | 1
  Dyspnea: Week 78 |  | 22.2 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Dyspnea: Post treatment efficacy visit 1: number analyzed (Participants) | 2 | 3
  Dyspnea: Post treatment efficacy visit 1 | 16.7 (23.57) | 3.7 (16.97)
  Dyspnea: Post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  Dyspnea: Post treatment efficacy visit 2 | -3.7 (44.91) | 22.2 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Dyspnea: Post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  Dyspnea: Post treatment efficacy visit 3 |  | 16.7 (7.86)
  Dyspnea: Post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  Dyspnea: Post treatment efficacy visit 5 |  | -11.1 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Dyspnea: 7 days post disease progression: number analyzed (Participants) | 31 | 29
  Dyspnea: 7 days post disease progression | 5.0 (17.88) | 2.3 (20.22)
  Dyspnea: 28 days post disease progression: number analyzed (Participants) | 18 | 16
  Dyspnea: 28 days post disease progression | 3.7 (16.61) | 10.4 (19.23)

12. Secondary Outcome: Randomized Part: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Health State Scores
Description: The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of these dimensions, the participant self-assigned a score: from 1 (no problems) to 5 (extreme problems). The 5 digit health states obtained for each dimension was converted into a single mean index value based on the EQ-5D crosswalk value set for the UK using the time trade-off method. This index ranges from -0.594 (worst health) to 1.0 (best health). A positive change from baseline indicates improvement. For subjects who discontinued treatment without disease progression, post-treatment efficacy visits 1, 2, 3 and 5 were conducted every 6 weeks (for the first 12 months since start of treatment) and every 12 weeks (after 12 months since start of treatment) until disease progression
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 120 | 117
Score on a scale
  Week 3: number analyzed (Participants) | 90 | 99
  Week 3 | -0.017 (0.1960) | -0.007 (0.1731)
  Week 6: number analyzed (Participants) | 77 | 86
  Week 6 | -0.016 (0.1972) | 0.001 (0.2283)
  Week 9: number analyzed (Participants) | 64 | 70
  Week 9 | -0.006 (0.1759) | 0.011 (0.1865)
  Week 12: number analyzed (Participants) | 61 | 59
  Week 12 | -0.028 (0.1849) | 0.014 (0.2315)
  Week 15: number analyzed (Participants) | 50 | 49
  Week 15 | -0.057 (0.2229) | -0.042 (0.1827)
  Week 18: number analyzed (Participants) | 51 | 48
  Week 18 | -0.062 (0.1835) | 0.009 (0.2810)
  Week 21: number analyzed (Participants) | 40 | 38
  Week 21 | -0.097 (0.2234) | 0.005 (0.1952)
  Week 24: number analyzed (Participants) | 35 | 34
  Week 24 | -0.070 (0.2075) | 0.027 (0.1900)
  Week 27: number analyzed (Participants) | 23 | 27
  Week 27 | -0.043 (0.1820) | 0.008 (0.2272)
  Week 30: number analyzed (Participants) | 18 | 25
  Week 30 | -0.023 (0.2378) | -0.014 (0.2068)
  Week 33: number analyzed (Participants) | 13 | 19
  Week 33 | -0.031 (0.2148) | 0.029 (0.2361)
  Week 36: number analyzed (Participants) | 12 | 15
  Week 36 | 0.017 (0.1942) | 0.050 (0.2743)
  Week 39: number analyzed (Participants) | 10 | 14
  Week 39 | -0.007 (0.1898) | -0.012 (0.2842)
  Week 42: number analyzed (Participants) | 10 | 15
  Week 42 | -0.010 (0.2286) | 0.116 (0.2180)
  Week 45: number analyzed (Participants) | 7 | 12
  Week 45 | 0.017 (0.1866) | -0.036 (0.1801)
  Week 48: number analyzed (Participants) | 6 | 9
  Week 48 | -0.087 (0.3178) | 0.003 (0.2424)
  Week 51: number analyzed (Participants) | 6 | 10
  Week 51 | -0.151 (0.2663) | 0.071 (0.2197)
  Week 54: number analyzed (Participants) | 6 | 7
  Week 54 | -0.102 (0.3527) | 0.056 (0.2011)
  Week 57: number analyzed (Participants) | 4 | 5
  Week 57 | 0.476 (0.2190) | 0.652 (0.1308)
  Week 60: number analyzed (Participants) | 3 | 4
  Week 60 | -0.193 (0.3653) | 0.149 (0.1616)
  Week 63: number analyzed (Participants) | 3 | 3
  Week 63 | -0.140 (0.3435) | 0.165 (0.1717)
  Week 66: number analyzed (Participants) | 2 | 2
  Week 66 | 0.034 (0.0481) | 0.124 (0.0085)
  Week 69: number analyzed (Participants) | 1 | 2
  Week 69 | 0.000 (NA) — NA: The standard deviation was not estimable as there was only one participant. | 0.340 (0.1230)
  Week 72: number analyzed (Participants) | 0 | 2
  Week 72 |  | 0.168 (0.0530)
  Week 75: number analyzed (Participants) | 0 | 1
  Week 75 |  | 0.130 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Week 78: number analyzed (Participants) | 0 | 1
  Week 78 |  | 0.130 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Post treatment efficacy visit 1: number analyzed (Participants) | 2 | 2
  Post treatment efficacy visit 1 | 0.100 (0.0955) | -0.026 (0.0368)
  Post treatment efficacy visit 2: number analyzed (Participants) | 3 | 1
  Post treatment efficacy visit 2 | 0.644 (0.1749) | 0.704 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Post treatment efficacy visit 3: number analyzed (Participants) | 0 | 2
  Post treatment efficacy visit 3 |  | 0.601 (0.0990)
  Post treatment efficacy visit 5: number analyzed (Participants) | 0 | 1
  Post treatment efficacy visit 5 |  | 1.000 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  7 days post disease progression: number analyzed (Participants) | 30 | 29
  7 days post disease progression | 0.639 (0.2558) | 0.657 (0.2654)
  28 days post disease progression: number analyzed (Participants) | 18 | 17
  28 days post disease progression | 0.692 (0.1633) | 0.692 (0.2149)

13. Secondary Outcome: Safety run-in Part: Maximum Plasma Concentration (Cmax) of Canakinumab
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Cmax of canakinumab was calculated from canakinumab plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Cycle 1 Day 1 at pre-dose and end of infusion and 24, 48, 168 and 336 hours (h) post-infusion. Each cycle is 21 days
Population: Canakinumab pharmacokinetic analysis set (PAS) in safety run-in part: all subjects who received at least one dose of canakinumab in the safety run-in part and have at least one evaluable canakinumab pharmacokinetic (PK) concentration. Only participants with an evaluable PK sample collected at each timepoint were included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 6
microgram/milliliter (ug/mL) | 13.4 (29.9)

14. Secondary Outcome: Safety run-in Part: Time of Maximum Plasma Concentration (Tmax) of Canakinumab
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Tmax of canakinumab was calculated from canakinumab plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
  Actual recorded sampling times were considered for the calculations.
Time Frame: Cycle 1 Day 1 at pre-dose and end of infusion and 24, 48, 168 and 336 hours (h) post-infusion. Each cycle is 21 days
Population: Canakinumab PAS in safety run-in part: all subjects who received at least one dose of canakinumab in the safety run-in part and have at least one evaluable canakinumab PK concentration. Only participants with an evaluable PK sample collected at each timepoint were included in this analysis
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 6
Hours (h) | 169 [48.2 to 336]

15. Secondary Outcome: Safety run-in Part: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of Canakinumab
Description: Venous whole blood samples were collected for pharmacokinetics characterization. AUClast of canakinumab was calculated from canakinumab plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Cycle 1 Day 1 at pre-dose and end of infusion and 24, 48, 168 and 336 hours (h) post-infusion. Each cycle is 21 days
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/mililiter (hr*ug/mL)
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 6
hour*microgram/mililiter (hr*ug/mL) | 5470 (30.5)

16. Secondary Outcome: Safety run-in Part: Cmax of Docetaxel
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Cmax of docetaxel was calculated from docetaxel plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at pre-infusion, end of infusion, and 2, 4, 6 and 8 hours post-dose. Each cycle is 21 days
Population: Docetaxel PAS in safety run-in part: all subjects who received at least one dose of canakinumab in the safety run-in part and have at least one evaluable docetaxel PK concentration. Number analyzed represents participants evaluable at specified time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/miliLiter (ng/mL)
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 8
nanogram/miliLiter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 7
  Cycle 1 Day 1 | 476 (182.5)
  Cycle 2 Day 1: number analyzed (Participants) | 5
  Cycle 2 Day 1 | 1630 (117.2)

17. Secondary Outcome: Safety run-in Part: Tmax of Docetaxel
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Tmax of docetaxel was calculated from docetaxel plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
  Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 8
Hour (hr)
  Cycle 1 Day 1: number analyzed (Participants) | 7
  Cycle 1 Day 1 | 1.08 [0.917 to 6.12]
  Cycle 2 Day 1: number analyzed (Participants) | 5
  Cycle 2 Day 1 | 1.00 [0.917 to 1.00]

18. Secondary Outcome: Safety run-in Part: AUClast of Docetaxel
Description: Venous whole blood samples were collected for pharmacokinetics characterization. AUClast of docetaxel was calculated from docetaxel plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour *nanogram/miliLiter (hr*ng/mL)
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel
Number analyzed (Participants) | 8
Hour *nanogram/miliLiter (hr*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 7
  Cycle 1 Day 1 | 884 (70.8)
  Cycle 2 Day 1: number analyzed (Participants) | 5
  Cycle 2 Day 1 | 2120 (86.5)

19. Secondary Outcome: Randomized Part: Pre-dose Plasma Trough Concentration (CTrough) of Canakinumab
Description: Venous whole blood samples were collected for pharmacokinetics characterization. CTrough of canakinumab was calculated from canakinumab plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Pre-dose on Cycle 1 Day 1, Cycle 4 Day 1, Cycle 6 Day 1, Cycle 12 Day 1 and Cycle 18 Day 1. Each cycle is 21 days.
Population: Canakinumab PAS in randomized part: all subjects who received at least one dose of canakinumab in the randomized part and have at least one evaluable canakinumab pharmacokinetic (PK) concentration. Number analyzed represents participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/miliLiter (ug/mL)
Arm/Group | Randomized Part: Canakinumab + Docetaxel
Number analyzed (Participants) | 112
microgram/miliLiter (ug/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 102
  Cycle 1 Day 1 | 0 (0)
  Cycle 4 Day 1: number analyzed (Participants) | 50
  Cycle 4 Day 1 | 20.5 (36.6)
  Cycle 6 Day 1: number analyzed (Participants) | 37
  Cycle 6 Day 1 | 23.7 (32.3)
  Cycle 12 Day 1: number analyzed (Participants) | 9
  Cycle 12 Day 1 | 25.6 (56.7)
  Cycle 18 Day 1: number analyzed (Participants) | 2
  Cycle 18 Day 1 | 28.3 (118.0)

20. Secondary Outcome: Randomized Part: Cmax of Docetaxel
Description: as for outcome 16
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 at pre-infusion, end of infusion, and 2, 4 and 6 hours post-dose. Each cycle is 21 days
Population: Docetaxel PAS in randomized part: all subjects who received at least one dose of canakinumab in the randomized part and have at least one evaluable docetaxel PK concentration. Number analyzed represents participants evaluable at specified time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/miliLiter (ng/mL)
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 26 | 23
nanogram/miliLiter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 26 | 22
  Cycle 1 Day 1 | 1570 (116.3) | 1190 (265.3)
  Cycle 4 Day 1: number analyzed (Participants) | 9 | 9
  Cycle 4 Day 1 | 1530 (118.7) | 940 (215.8)

21. Secondary Outcome: Randomized Part: Tmax of Docetaxel
Description: as for outcome 17
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 at pre-infusion, end of infusion, and 2, 4 and 6 hours post-dose. Each cycle is 21 days
Population: as for outcome 20
Measure: Median (Full Range); unit: Hour
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 26 | 23
Hour
  Cycle 1 Day 1: number analyzed (Participants) | 26 | 22
  Cycle 1 Day 1 | 1.09 [0.517 to 5.83] | 1.10 [0.933 to 6.08]
  Cycle 4 Day 1: number analyzed (Participants) | 9 | 9
  Cycle 4 Day 1 | 1.15 [0.0833 to 3.83] | 1.08 [1.00 to 1.42]

22. Secondary Outcome: Randomized Part: AUClast of Docetaxel
Description: as for outcome 18
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 at pre-infusion, end of infusion, and 2, 4 and 6 hours post-dose. Each cycle is 21 days
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/miliLiter (h*ng/mL)
Arm/Group | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 22 | 19
hour*nanogram/miliLiter (h*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 19 | 17
  Cycle 1 Day 1 | 2530 (79.3) | 1790 (157.4)
  Cycle 4 Day 1: number analyzed (Participants) | 7 | 8
  Cycle 4 Day 1 | 2210 (66.4) | 1530 (130.9)

23. Secondary Outcome: Randomized Part: Canakinumab Antidrug Antibodies (ADA) at Baseline
Description: ADA prevalence at baseline was calculated as the percentage of participants who had an ADA positive result at baseline
Time Frame: Baseline
Population: All participants randomized to canakinumab+docetaxel arm
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Part: Canakinumab + Docetaxel
Number analyzed (Participants) | 120
Participants | 1

24. Secondary Outcome: Randomized Part: Canakinumab ADA Incidence On-treatment
Description: ADA incidence on-treatment was calculated as the percentage of participants who were treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: Pre-dose at Cycle 1 Day 1, Cycle 4 Day 1, Cycle 6 Day 1, Cycle 12 Day 1 , end of treatment, and 130 days after end of treatment through final analysis data cutoff date of 08-Jan-2021 (assessed up to 18 months). Each cycle is 21 days
Population: All participants randomized to canakinumab+docetaxel arm
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Part: Canakinumab + Docetaxel
Number analyzed (Participants) | 120
Participants | 0

25. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from screening to the first day of treatment, for a maximum duration of 28 days.
  On-treatment deaths due to any cause were collected from first dose of study treatment to 130 days after the last dose of study treatment.
  Post-treatment survival follow-up deaths were collected from day 131 after last dose of study treatment to end of study.
  All deaths refer to the sum of pre-treatment, on-treatment and post-treatment deaths.
Time Frame: Pre-treatment: up to 28 days before Day 1;On-treatment: up to approximately 10 months (safety run-in) or 25 months (randomized); post-treatment survival follow-up deaths: Up to approximately 16 months (safety run in) or 25 months (randomized)
Population: Safety run-in part: FAS including all subjects to whom study treatment was assigned.
  Randomized part: FAS including all participants to whom study treatment was assigned by randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Safety run-in Part: Canakinumab+Docetaxel | Randomized Part: Canakinumab + Docetaxel | Randomized Part: Placebo + Docetaxel
Number analyzed (Participants) | 8 | 120 | 117
Participants
  Pre-treatment deaths | 0 | 0 | 1
  On-treatment deaths: number analyzed (Participants) | 8 | 120 | 114
  On-treatment deaths | 6 | 45 | 37
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 2 | 75 | 77
  Post-treatment survival follow-up deaths | 2 | 40 | 38
  All deaths | 8 | 85 | 76

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse events (AEs) were collected from first administration of study treatment to 130 days after date of last administration, up to approximately 10 months (safety run-in) or 25 months (randomized). Deaths were collected from day of subject's informed consent until end of study, up to approximately 16 months (safety run in) or 25 months (randomized)
Description: Treatment-emergent AEs refer to any signs or symptoms observed during the study treatment and up to 130 days after treatment, considering the Safety Set. This set includes all subjects who were assigned study treatment and received at least one dose, including incomplete infusions.
  All-Cause Mortality analysis encompasses the Full Analysis Set, including all subjects who were assigned study treatment
Groups:
- All Participants (Pre-treatment): Deaths were collected in the pre-treatment period (from day of patient's informed consent to the day before first administration of study treatment )
- Safety run-in Part: Canakinumab+Docetaxel (On-treatment): AEs during on-treatment period (up to 130 days post-treatment)
- Safety run-in Part: Canakinumab+Docetaxel (Post-treatment Follow-up); Randomized Part: Placebo + Docetaxel (Post-treatment Follow-up): Deaths collected in the post- treatment follow-up period (starting from day 131 post- treatment). No AEs were collected during this period
- Randomized Part: Canakinumab + Docetaxel (On-treatment); Randomized Part: Placebo + Docetaxel (On-treatment): AEs during on-treatment period (up to 30 days post-treatment)
- Randomized Part: Canakinumab + Docetaxel (Post-treatment Follow-up): Deaths collected in the post- treatment follow-up period (starting from day 131 post-treatment). No AEs were collected during this period
Arm/Group | All Participants (Pre-treatment) | Safety run-in Part: Canakinumab+Docetaxel (On-treatment) | Safety run-in Part: Canakinumab+Docetaxel (Post-treatment Follow-up) | Randomized Part: Canakinumab + Docetaxel (On-treatment) | Randomized Part: Canakinumab + Docetaxel (Post-treatment Follow-up) | Randomized Part: Placebo + Docetaxel (On-treatment) | Randomized Part: Placebo + Docetaxel (Post-treatment Follow-up)
All-Cause Mortality (participants affected / at risk) | 1/245 | 6/8 | 2/2 | 45/120 | 40/75 | 37/114 | 38/77
Serious Adverse Events (participants affected / at risk) | 0/0 | 6/8 | 0/0 | 55/120 | 0/0 | 50/114 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 7/8 | 0/0 | 111/120 | 0/0 | 109/114 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Pre-treatment) (N=0) | Safety run-in Part: Canakinumab+Docetaxel (On-treatment) (N=8) | Safety run-in Part: Canakinumab+Docetaxel (Post-treatment Follow-up) (N=0) | Randomized Part: Canakinumab + Docetaxel (On-treatment) (N=120) | Randomized Part: Canakinumab + Docetaxel (Post-treatment Follow-up) (N=0) | Randomized Part: Placebo + Docetaxel (On-treatment) (N=114) | Randomized Part: Placebo + Docetaxel (Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 0 | NA | 6 | NA | 8 | NA
Leukopenia (Blood and lymphatic system disorders) | NA | 0 | NA | 1 | NA | 1 | NA
Neutropenia (Blood and lymphatic system disorders) | NA | 1 | NA | 4 | NA | 5 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Atrial fibrillation (Cardiac disorders) | NA | 0 | NA | 2 | NA | 1 | NA
Cardiac tamponade (Cardiac disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Cardio-respiratory arrest (Cardiac disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Pericardial effusion (Cardiac disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Hypopituitarism (Endocrine disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Abdominal pain (Gastrointestinal disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Abdominal pain upper (Gastrointestinal disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Colitis ulcerative (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Diarrhoea (Gastrointestinal disorders) | NA | 0 | NA | 2 | NA | 2 | NA
Dysphagia (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Ileus (Gastrointestinal disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Nausea (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Small intestine ulcer (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Stomatitis (Gastrointestinal disorders) | NA | 0 | NA | 0 | NA | 2 | NA
Vomiting (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Asthenia (General disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Chest pain (General disorders) | NA | 0 | NA | 2 | NA | 0 | NA
Disease progression (General disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Fatigue (General disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Generalised oedema (General disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Malaise (General disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Mucosal inflammation (General disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Oedema peripheral (General disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Pyrexia (General disorders) | NA | 0 | NA | 6 | NA | 2 | NA
Abdominal sepsis (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Bacteraemia (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Bacterial infection (Infections and infestations) | NA | 1 | NA | 0 | NA | 0 | NA
Bronchitis (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
COVID-19 (Infections and infestations) | NA | 0 | NA | 1 | NA | 1 | NA
COVID-19 pneumonia (Infections and infestations) | NA | 0 | NA | 1 | NA | 1 | NA
Clostridium difficile colitis (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Device related infection (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Diverticulitis (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Erysipelas (Infections and infestations) | NA | 0 | NA | 1 | NA | 1 | NA
Escherichia sepsis (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Escherichia urinary tract infection (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Febrile infection (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Gastroenteritis (Infections and infestations) | NA | 0 | NA | 1 | NA | 1 | NA
Gastroenteritis viral (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Infection (Infections and infestations) | NA | 0 | NA | 1 | NA | 1 | NA
Infectious pleural effusion (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Influenza (Infections and infestations) | NA | 1 | NA | 0 | NA | 0 | NA
Lower respiratory tract infection (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Neutropenic sepsis (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Pneumonia (Infections and infestations) | NA | 2 | NA | 13 | NA | 8 | NA
Pneumonia pneumococcal (Infections and infestations) | NA | 1 | NA | 0 | NA | 0 | NA
Pneumonia pseudomonal (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Post procedural sepsis (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Pulmonary sepsis (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Respiratory tract infection (Infections and infestations) | NA | 0 | NA | 3 | NA | 4 | NA
Sepsis (Infections and infestations) | NA | 0 | NA | 2 | NA | 1 | NA
Septic shock (Infections and infestations) | NA | 0 | NA | 3 | NA | 1 | NA
Spinal cord infection (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Upper respiratory tract infection (Infections and infestations) | NA | 0 | NA | 1 | NA | 0 | NA
Urinary tract infection (Infections and infestations) | NA | 0 | NA | 0 | NA | 4 | NA
Urosepsis (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Vulvovaginitis (Infections and infestations) | NA | 0 | NA | 0 | NA | 1 | NA
Femur fracture (Injury, poisoning and procedural complications) | NA | 1 | NA | 0 | NA | 0 | NA
Hip fracture (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | NA | 0 | NA
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | NA | 0 | NA | 0 | NA | 1 | NA
Procedural pneumothorax (Injury, poisoning and procedural complications) | NA | 0 | NA | 0 | NA | 1 | NA
Aspartate aminotransferase increased (Investigations) | NA | 0 | NA | 0 | NA | 1 | NA
Gamma-glutamyltransferase increased (Investigations) | NA | 0 | NA | 0 | NA | 1 | NA
Neutrophil count decreased (Investigations) | NA | 0 | NA | 1 | NA | 1 | NA
White blood cell count decreased (Investigations) | NA | 0 | NA | 1 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Dehydration (Metabolism and nutrition disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 0 | NA | 3 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 0 | NA | 2 | NA
Fistula (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 0 | NA | 1 | NA
Cerebrovascular accident (Nervous system disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Dizziness (Nervous system disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Ischaemic stroke (Nervous system disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Monoplegia (Nervous system disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Syncope (Nervous system disorders) | NA | 0 | NA | 1 | NA | 1 | NA
Acute kidney injury (Renal and urinary disorders) | NA | 0 | NA | 2 | NA | 0 | NA
Balanoposthitis (Reproductive system and breast disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 4 | NA | 5 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 3 | NA | 1 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 2 | NA | 0 | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 2 | NA | 1 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | NA | 3 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 3 | NA | 1 | NA
Aneurysm (Vascular disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Haematoma (Vascular disorders) | NA | 0 | NA | 0 | NA | 1 | NA
Hypotension (Vascular disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Superior vena cava syndrome (Vascular disorders) | NA | 0 | NA | 1 | NA | 0 | NA
Thrombosis (Vascular disorders) | NA | 0 | NA | 1 | NA | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Pre-treatment) (N=0) | Safety run-in Part: Canakinumab+Docetaxel (On-treatment) (N=8) | Safety run-in Part: Canakinumab+Docetaxel (Post-treatment Follow-up) (N=0) | Randomized Part: Canakinumab + Docetaxel (On-treatment) (N=120) | Randomized Part: Canakinumab + Docetaxel (Post-treatment Follow-up) (N=0) | Randomized Part: Placebo + Docetaxel (On-treatment) (N=114) | Randomized Part: Placebo + Docetaxel (Post-treatment Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | NA | 1 | NA | 32 | NA | 33 | NA
Leukopenia (Blood and lymphatic system disorders) | NA | 1 | NA | 6 | NA | 15 | NA
Neutropenia (Blood and lymphatic system disorders) | NA | 2 | NA | 22 | NA | 25 | NA
Atrial fibrillation (Cardiac disorders) | NA | 1 | NA | 0 | NA | 0 | NA
Tachycardia (Cardiac disorders) | NA | 1 | NA | 1 | NA | 2 | NA
Cushingoid (Endocrine disorders) | NA | 1 | NA | 0 | NA | 0 | NA
Abdominal pain (Gastrointestinal disorders) | NA | 1 | NA | 7 | NA | 4 | NA
Constipation (Gastrointestinal disorders) | NA | 0 | NA | 22 | NA | 24 | NA
Diarrhoea (Gastrointestinal disorders) | NA | 3 | NA | 41 | NA | 31 | NA
Dyspepsia (Gastrointestinal disorders) | NA | 0 | NA | 7 | NA | 0 | NA
Nausea (Gastrointestinal disorders) | NA | 1 | NA | 28 | NA | 29 | NA
Odynophagia (Gastrointestinal disorders) | NA | 1 | NA | 1 | NA | 1 | NA
Stomatitis (Gastrointestinal disorders) | NA | 0 | NA | 9 | NA | 6 | NA
Vomiting (Gastrointestinal disorders) | NA | 2 | NA | 15 | NA | 14 | NA
Asthenia (General disorders) | NA | 2 | NA | 28 | NA | 37 | NA
Chest pain (General disorders) | NA | 0 | NA | 5 | NA | 10 | NA
Fatigue (General disorders) | NA | 1 | NA | 33 | NA | 19 | NA
Influenza like illness (General disorders) | NA | 1 | NA | 1 | NA | 3 | NA
Malaise (General disorders) | NA | 0 | NA | 7 | NA | 7 | NA
Mucosal inflammation (General disorders) | NA | 0 | NA | 4 | NA | 12 | NA
Oedema (General disorders) | NA | 1 | NA | 5 | NA | 2 | NA
Oedema peripheral (General disorders) | NA | 3 | NA | 22 | NA | 25 | NA
Pyrexia (General disorders) | NA | 1 | NA | 14 | NA | 18 | NA
Bronchitis (Infections and infestations) | NA | 1 | NA | 4 | NA | 3 | NA
Folliculitis (Infections and infestations) | NA | 1 | NA | 0 | NA | 1 | NA
Nasopharyngitis (Infections and infestations) | NA | 1 | NA | 5 | NA | 2 | NA
Pneumonia (Infections and infestations) | NA | 0 | NA | 7 | NA | 4 | NA
Respiratory tract infection (Infections and infestations) | NA | 1 | NA | 7 | NA | 3 | NA
Upper respiratory tract infection (Infections and infestations) | NA | 0 | NA | 5 | NA | 6 | NA
Urinary tract infection (Infections and infestations) | NA | 0 | NA | 8 | NA | 7 | NA
Alanine aminotransferase increased (Investigations) | NA | 0 | NA | 7 | NA | 3 | NA
Aspartate aminotransferase increased (Investigations) | NA | 0 | NA | 7 | NA | 0 | NA
Gamma-glutamyltransferase increased (Investigations) | NA | 2 | NA | 5 | NA | 6 | NA
Haemoglobin decreased (Investigations) | NA | 1 | NA | 1 | NA | 2 | NA
Neutrophil count decreased (Investigations) | NA | 0 | NA | 17 | NA | 11 | NA
SARS-CoV-2 test negative (Investigations) | NA | 0 | NA | 10 | NA | 13 | NA
Weight decreased (Investigations) | NA | 1 | NA | 9 | NA | 8 | NA
White blood cell count decreased (Investigations) | NA | 2 | NA | 12 | NA | 8 | NA
Decreased appetite (Metabolism and nutrition disorders) | NA | 0 | NA | 32 | NA | 31 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | NA | 0 | NA | 7 | NA | 5 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | NA | 0 | NA | 8 | NA | 7 | NA
Hyponatraemia (Metabolism and nutrition disorders) | NA | 0 | NA | 7 | NA | 7 | NA
Steroid diabetes (Metabolism and nutrition disorders) | NA | 1 | NA | 0 | NA | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 11 | NA | 10 | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | 1 | NA | 8 | NA | 6 | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | NA | 1 | NA | 0 | NA | 0 | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 1 | NA | 6 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 9 | NA | 9 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 6 | NA | 7 | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 0 | NA | 2 | NA
Dysgeusia (Nervous system disorders) | NA | 0 | NA | 8 | NA | 3 | NA
Headache (Nervous system disorders) | NA | 0 | NA | 8 | NA | 6 | NA
Neuropathy peripheral (Nervous system disorders) | NA | 1 | NA | 9 | NA | 15 | NA
Paraesthesia (Nervous system disorders) | NA | 0 | NA | 12 | NA | 8 | NA
Taste disorder (Nervous system disorders) | NA | 1 | NA | 1 | NA | 0 | NA
Anxiety (Psychiatric disorders) | NA | 1 | NA | 5 | NA | 2 | NA
Insomnia (Psychiatric disorders) | NA | 1 | NA | 7 | NA | 8 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 2 | NA | 16 | NA | 19 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 2 | NA | 27 | NA | 26 | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 3 | NA | 5 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 5 | NA | 6 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 10 | NA | 10 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 4 | NA | 6 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 6 | NA | 3 | NA
Alopecia (Skin and subcutaneous tissue disorders) | NA | 1 | NA | 31 | NA | 44 | NA
Dry skin (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 4 | NA | 7 | NA
Nail disorder (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 7 | NA | 8 | NA
Night sweats (Skin and subcutaneous tissue disorders) | NA | 1 | NA | 0 | NA | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 10 | NA | 9 | NA
Psoriasis (Skin and subcutaneous tissue disorders) | NA | 1 | NA | 0 | NA | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 12 | NA | 10 | NA
Hypotension (Vascular disorders) | NA | 1 | NA | 6 | NA | 5 | NA
Phlebitis (Vascular disorders) | NA | 1 | NA | 0 | NA | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03626545/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03626545/SAP_001.pdf